CLINICAL TRIAL: NCT04275310
Title: Microeconomic Intervention to Reduce HIV Transmission in Economically Disadvantaged Transgender Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of funding
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HM20011245; R34MH115775 (NIH)
Record Dates: First submitted 2020-02-12; First posted 2020-02-19 (Actual); Results first posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Hiv; Transgenderism
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Transsexualism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microeconomic intervention (Experimental)
  Interventions: Behavioral: Microeconomic Intervention
- Waitlisted control (No Intervention)

INTERVENTIONS:
Behavioral: Microeconomic Intervention — The intervention will consist of six sessions on six different days. Sessions will be held at VCU or at one of VCU's community partners. Each session will last for around 2 ½ hours (around 15 hours total). There will be breaks and food will be provided. During the sessions the facilitators will provide education on a variety of topics, including economic services that are available to people living in Richmond, job skills (such as creating a resume and dealing with discrimination at work), personal finance education, gender transition ideas, and HIV prevention. The sessions will occur in a group of about 4-10 transgender women.
  Arms: Microeconomic intervention

SUMMARY:
The purpose of this research study is to learn more about the economic situations, discrimination experiences, and risk behaviors of transgender women. The ultimate purpose of the study is to test an intervention to improve financial conditions and reduce HIV risk behaviors in transgender women.

DETAILED DESCRIPTION:
The study includes a microeconomic intervention which will provide education on a variety of economic and behavioral topics. Participants will complete questionnaires on multiple occasions during the study.

ELIGIBILITY:
Inclusion Criteria:

* Transgender woman
* 18-45 years of age

At least one of the following economic vulnerability factors:

unemployment or underemployment [less than 20 hours/week], low income [less than the Medicaid poverty threshold], housing insecurity in the past year or food insecurity in the past year

• Behavioral vulnerability to HIV transmission (reported at least one episode of unprotected sex in prior 6 months or at least one other behavioral HIV transmission risk factor in the past 6 months: [transactional sex, multiple sexual partners, 1-time sexual partner, sex under the influence of drugs or alcohol, sex with partner of unknown HIV status).

Exclusion Criteria:

* obvious signs of intoxication or cognitive impairment
* cannot speak English.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Transgender women
Enrollment: 4 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Benotsch, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Waitlisted Control: Overflow
Period: Overall Study
Arm/Group | Microeconomic Intervention | Waitlisted Control
Started | 4 | 0
Completed | 0 | 0
Not Completed | 4 | 0
Not completed — Non-randomized due to running out of funding | 4 | 0

BASELINE CHARACTERISTICS:
Population: No analysis was completed as no study procedures were ever initiated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Microeconomic Intervention | Waitlisted Control | Total
Number analyzed (Participants) | 4 | 0 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 0 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 0 | 4
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 |  | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Employment Status
Description: Number of participants whose status with respect to employment improves after the intervention.
Time Frame: Baseline to up to 9 months
Population: Analysis was not completed due to low enrollment, loss of funding and no participants completing study-related activities.
Arm/Group | Microeconomic Intervention | Waitlisted Control
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change in Income
Description: Number of participants whose income increases after the intervention.
Time Frame: Baseline to up to 9 months
Population: as for outcome 1
Arm/Group | Microeconomic Intervention | Waitlisted Control
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Change in Housing Stability
Description: Number of participants whose access to stable permanent housing improves after the intervention.
Time Frame: Baseline to up to 9 months
Population: as for outcome 1
Arm/Group | Microeconomic Intervention | Waitlisted Control
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Change in Savings
Description: Number of participants whose savings increase after the intervention.
Time Frame: Baseline to up to 9 months
Population: as for outcome 1
Arm/Group | Microeconomic Intervention | Waitlisted Control
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Change in Self Reported HIV Risk Behavior
Description: Number of participants whose self-reports of behaviors known to increase risk for HIV goes down after the intervention.
Time Frame: Baseline to up to 9 months
Population: as for outcome 1
Arm/Group | Microeconomic Intervention | Waitlisted Control
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Change in Compliance With Recommended Biomedical Prevention or Treatment
Description: Number of participants who demonstrate higher compliance with recommended biomedical prevention or treatment behaviors after the intervention.
Time Frame: Baseline to up to 9 months
Population: as for outcome 1
Arm/Group | Microeconomic Intervention | Waitlisted Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 months
Description: For the waitlisted control group, the number of participants at risk for serious adverse events, all-cause mortality and other adverse events is listed as "0." This is because no participants were enrolled into this group.
Arm/Group | Microeconomic Intervention | Waitlisted Control
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/0
Other Adverse Events (participants affected / at risk) | 0/4 | 0/0

LIMITATIONS AND CAVEATS:
Early termination due to loss of funding. As a result a small number of participants were consented. None of those consented did any study-related activities and therefore no data was collected to analyze.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/10/NCT04275310/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/10/NCT04275310/ICF_001.pdf